CLINICAL TRIAL: NCT01806441
Title: Impact of a Short-Term High Fat Diet Versus A Short-Term Low Fat Diet on Expression of the Key Intestinal Genes Involved in the Cholesterol and Fatty Acid Metabolism Pathways
Brief Title: Impact of a Short-Term High Fat or Low Fat Diet on Intestinal Genes Expression Involved in the Cholesterol and Fatty Acid Metabolism
Acronym: DGENES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Patrick Couture, MD, FRCP, PhD, Laval University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: INAF-125-05-06
Record Dates: First submitted 2013-03-04; First posted 2013-03-07 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Gene Expression
MeSH Terms: interventions — Diet, High-Fat; Diet, Fat-Restricted

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3-days high fat diet (Experimental): During 3 days, subjects eat a diet high in fat (percent of total caloric intake: 15.0% from proteins; 49,8% from carbohydrates; 37.0% from fat).
  Interventions: Other: 3-days high fat diet
- 3-days low fat diet (Active Comparator): During 3 days, subjects eat a diet low in fat (percent of caloric intake: 15.0% from proteins; 61,8% from carbohydrates; 25.0% from fats).
  Interventions: Other: 3-days low fat diet

INTERVENTIONS:
Other: 3-days high fat diet — During 3 days, subjects eat a diet high in fat (percent of total caloric intake: 15.0% from proteins; 49,8% from carbohydrates; 37.0% from fat).
  Arms: 3-days high fat diet
Other: 3-days low fat diet — During 3 days, subjects eat a diet low in fat (percent of caloric intake: 15.0% from proteins; 61,8% from carbohydrates; 25.0% from fats).
  Arms: 3-days low fat diet

SUMMARY:
Dietary fat has been shown to modulate cholesterol and fatty acids homeostasis and several lines of evidence suggest that this effect is associated with changes in the regulation of different genes at the intestine level involved in the cholesterol and fatty acid metabolism pathways. The present study will examine the impact of a short-term high fat diet versus a short-term low fat diet on expression of Niemann-Pick C1-like 1 (NPC1L1), adenosine triphosphate (ATP) binding cassette transporters (ABCG5/8), microsomal triglyceride transfer protein (MTP) and fatty acid transport protein-4 (FATP4), which have been shown to play a critical role in intestinal cholesterol absorption, chylomicron synthesis and dietary lipid absorption. Gene expression studies will be performed on duodenal biopsies. The primary hypothesis is that a short-term high fat diet will significantly decrease duodenal messenger ribonucleic acid (mRNA) levels of NPC1L1, ABCG5/8, MTP and FATP4 as compared with a short-term low fat diet.

ELIGIBILITY:
Inclusion Criteria:

* Males 18 to 50 years of age
* Non-smoker
* Body mass index between 20.0 and 30.0 kg/m2
* Plasma LDL-cholesterol levels between the 25th and 75th percentile for their age at day -14
* Plasma triglyceride levels < 1.7 mmol/L (150 mg/dl) at day -14
* Plasma HDL-cholesterol levels between 0.9 (35 mg/dl) and 1.6 mmol/L (60 mg/dl) at day -14
* Subjects must be willing to give written informed consent and able to adhere to the diet schedule and visit schedule
* Patients should be otherwise healthy, without elevations in hepatic transaminases or creatine kinase (CK) or abnormal renal function or coagulation

Exclusion Criteria:

* Patients with extreme dyslipidemias, such as familial hypercholesterolemia will be excluded
* Subjects will be excluded if they have cardiovascular disease (CHD, cerebrovascular disease or peripheral arterial disease) or if they are taking other medications known to affect lipoprotein metabolism (eg. steroids, beta blockers, thiazide diuretics, other lipid lowering agents, significant alcohol intake etc.)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-02; Primary Completion 2009-05 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Change in duodenal mRNA expression of NPC1L1, ABCG5/8, MTP and FATP4. | At the end of the two 3-days diets (day 3 and day 17).
  Six biopsies (3 X 3 mm) will be obtained from the second portion of the duodenum during gastro-duodenoscopy. Biopsy specimen will be stored at -86°C before mRNA extraction. Total RNA will be isolated and used for polymerase chain reaction (PCR) quantification.

SECONDARY OUTCOMES:
Change in surrogate markers of cholesterol absorption and synthesis. | At the end of the two 3-days diets (day 3 and day 17).

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Couture, MD,FRCP,PhD, Principal Investigator — Laval University
Locations (1):
- Institute of nutrition and functional food, Québec, Quebec, Canada

REFERENCES:
- [Derived] Tremblay AJ, Lamarche B, Guay V, Charest A, Lemelin V, Couture P. Short-term, high-fat diet increases the expression of key intestinal genes involved in lipoprotein metabolism in healthy men. Am J Clin Nutr. 2013 Jul;98(1):32-41. doi: 10.3945/ajcn.113.060251. Epub 2013 May 29. PMID 23719552